## STUDY TITLE:

INCIDENCE OF AND FACTORS ASSOCIATED WITH POST-OPERATIVE NAUSEA AND VOMITING FOLLOWING SURGERY UNDER REGIONAL ANAESTHESIA

**NCT NUMBER:** 

NCT03835234

**DOCUMENT DATE:** 

31/01/2019

 Table 1: Baseline characteristics of study participants

| | Post -operative Nausea<br>No [n=224,%] | P-value | |
|---|---|---|---|
| Demographic | | | |
| Urgency of surgery | | | 0.179 |
| Elective | 107 (58.2) | 77 (41.8) | |
| Emergency | 117 (65.0) | 63 (35.0) | |
| Sex | | | 0.650 |
| Male | 56 (59.6) | 38(40.4) | |
| Female | 168 (62.2) | 102(37.8) | |
| ASA classification | | | < 0.0011 |
| I | 26 (42.6) | 35 (57.4) | |
| II | 196 (66.2) | 100 (33.8) | |
| III | 2 (28.6) | 5 (71.4) | |
| Age; median (IQR) | 28 (23 - 37) | 30 (24 - 42) | 0.039a |
| Patient experience | , , , | | |
| Ever had nausea or | | | 0.013 |
| vomiting | | | |
| Yes | 154 (57.9) | 112 (42.1) | |
| No | 70 (72.2) | 27 (27.8) | |
| Description of | , , | , , | 0.110 |
| experience | | | |
| Very unfavorable | 14 (45.2) | 17 (54.8) | |
| Unfavorable | 84 (65.6) | 44 (34.4) | |
| Neutral | 106 (61.3) | 67 (38.7) | |
| Post-operative nausea and vomiting | | , , , | |
| History of PONV | | | < 0.001 |
| Yes | 23 (39.7) | 35 (60.3) | |
| No | 201 (65.7) | 105 (34.3) | |
| History of motion | | ( ) | 0.002 |
| sickness | | | ***** |
| Yes | 80 (52.3) | 73 (47.7) | |
| No | 144 (68.3) | 67 (31.7) | |
| Alcohol use | , | , , | 0.227 |
| Yes | 31 (54.4) | 26 (45.6) | |
| No | 193 (62.9) | 114 (37.1) | |
| Smoker | (**) | (5) | 0.7121 |
| Yes | 5 (71.4) | 2 (28.6) | <b></b> |
| No | 219 (61.5) | 137 (38.5) | |
| Time since last feed | 217 (01.0) | 20, (00.0) | 0.007 |
| (hours) | | | 0.007 |
| <u>≤2</u> | 27 (45.8) | 32 (54.2) | |
| <u>==</u><br>>2 | 197 (64.6) | 108 (35.4) | |
| Type of feeds | 157 (0110) | 100 (33.1) | 0.018 |
| Solids | 82 (67.2) | 40 (32.8) | 0.010 |
| Semi-solids | 57 (50.9) | 55 (49.1) | |
| Liquids | 85 (65.9) | 44 (34.1) | |
| Anesthesia provider | 05 (05.7) | TT (JT.1) | 0.2881 |
| <u>*</u> | 5 (92.2) | 1 (16.7) | U.400 |
| AO student trainee | 5 (83.3) | 1 (16.7) | |

| AO | 77 (56.6) | 59 (43.4) | |
|-------------------------------|------------|-----------|-------|
| SHO | 102 (63.0) | 60 (37.0) | |
| Anesthesiologist | 36 (69.2) | 16 (30.8) | |
| Length of the | | | |
| operation | | | |
| <b>Duration of anesthesia</b> | | | 0.770 |
| (minutes) | | | |
| 30 | 20 (64.5) | 11 (35.5) | |
| 30 – 60 | 109 (59.9) | 73 (40.1) | |
| 60 – 120 | 73 (64.6) | 40 (35.4) | |
| >120 | 21 (56.8) | 16 (43.2) | |
| <b>Duration of surgery</b> | | | 0.867 |
| (minutes) | | | |
| 30 | 24 (64.9) | 13 (35.1) | |
| 30 – 60 | 119 (61.3) | 75 (38.7) | |
| 60 – 120 | 59 (62.1) | 36 (37.9) | |
| >120 | 20 (55.6) | 16 (44.4) | |
| | | , , , | |

Figure 1: Incidence of postoperative nausea and vomiting in patients having surgery under regional anaesthesia at Mulago hospital



The incidence of postoperative nausea and vomiting in patients who had surgery under regional anaesthesia at Mulago hospital was found to be 38%.

Table 2: Bivariate analysis for risk factors for  ${\bf PONV}$ 

| Characteristics | PONV | P-value | |
|---|---|---|---|
| | No (n=224, %) | Yes (n=140, %) | |
| Urgency of surgery | | == ((1, 0) | 0.179 |
| Elective | 107 (58.2) | 77 (41.8) | |
| Emergency | 117 (65.0) | 63 (35.0) | |
| Sex | | | 0.650 |
| Male | 56 (59.6) | 38 (40.4) | |
| Female | 168 (62.2) | 102 (37.8) | |
| ASA classification | | | <0.0011 |
| 1 | 26 (42.6) | 35 (57.4) | |
| 2 | 196 (66.2) | 100 (33.8) | |
| 3 | 2 (28.6) | 5 (71.4) | |
| Age ; median (IQR) | 28 (23 - 37) | 30 (24 - 42) | 0.039 <sup>a</sup> |
| History of PONV | 23 (39.7) | 35 (60.3) | < 0.001 |
| History of motion sickness | 80 (52.3) | 73 (47.7) | 0.002 |
| Alcohol use | 31 (54.4) | 26 (45.6) | 0.227 |
| Non Smoker | 219 (61.5) | 137 (38.5) | 0.7121 |
| Time since last feed (hours) | | | 0.007 |
| ≤2 | 27 (45.8) | 32 (54.2) | |
| >2 | 197 (64.6) | 108 (35.4) | |
| Type of feeds | | | 0.018 |
| Solids | 82 (67.2) | 40 (32.8) | |
| Semi-solids | 57 (50.9) | 55 (49.1) | |
| Liquids | 85 (65.9) | 44 (34.1) | |
| Duration of surgery (minutes) | , , | , , | 0.867 |
| 30 | 24 (64.9) | 13 (35.1) | |
| 30 - 60 | 119 (61.3) | 75 (38.7) | |
| 60 - 120 | 59 (62.1) | 36 (37.9) | |
| >120 | 20 (55.6) | 16 (44.4) | |
| Drugs used during anesthesia | | | |
| Opioids State of the control of the | 114 (67.1) | 56 (32.9) | 0.056 |
| Anti-emetics | 49 (53.3) | 43 (46.7) | 0.062 |
| Sedatives | , (55.5) | 19 (32.2) | 0.285 |
| SBP | | (- ) | 0.0011 |
| <110 | 121 (65.4) | 64 (34.6) | - • • • • |
| <90 | 45 (44.6) | 56 (55.4) | |
| <50 | 1 (0.6) | 0 (0.0) | |
| DBP | 1 (0.0) | 3 (0.0) | 0.097 |
| <90 | 26 (76.5) | 8 (23.5) | 0.071 |
| <70 | 113 (60.1) | 75 (39.9) | |
| <50 | 66 (55.9) | 52 (44.1) | |
| Post-operative opioids received | 30 (33.5) | 22 (11.1) | 0.800 |
| Yes | 136 (61.0) | 87 (39.0) | 0.000 |
| No | 86 (62.3) | 52 (37.7) | |

P- chi-square p-values, P¹- fishers exact p-values, Pª- Rank sum p-values

Table 3: Multivariable logistic regression model showing factors associated with Post-operative nausea and vomiting

| Characteristics | Unadjusted | P-value | Adjusted | P-value |
|---|---|---|---|---|
| | Odds ratio (95% CI) | | Odds ratio (95% CI) | |
| Age | 1.03 (1.01 - 1.04) | 0.003 | 1.03 (1.01 - 1.06) | 0.011 |
| Urgency | | | | |
| Elective | 1.00 | | 1.00 | |
| Emergency | 0.75 (0.49 - 1.14) | 0.180 | 1.68 (0.82 - 3.44) | 0.153 |
| ASA classification | | | | |
| 1 | 1.00 | | 1.00 | |
| 2 | 0.38 (0.22 - 0.66) | 0.001 | 0.36 (0.16 - 0.83) | 0.016 |
| 3 | 1.86 (0.33 - 10.34) | 0.480 | 1.38 (0.17 - 11.32) | 0.763 |
| History of PONV | | | | |
| No | 1.00 | | 1.00 | |
| Yes | 2.91 (1.64 - 5.19) | < 0.001 | 2.61 (1.25 - 5.46) | 0.011 |
| History of motion sickness | | | | |
| No | 1.00 | | 1.00 | |
| Yes | 1.96 (1.28 - 3.01) | 0.002 | 2.36 (1.20 - 4.65) | 0.013 |
| Ever had nausea or | | | | |
| vomiting | | | | |
| No | 1.00 | | 1.00 | |
| Yes | 1.89 (1.14 - 3.13) | 0.014 | 3.49 (1.53 - 7.96) | 0.003 |
| Time since last feed | | | | |
| (hours) | | | | |
| >2 | 1.00 | | 1.00 | |
| ≤2 | 2.16 (1.23 - 3.80) | 0.007 | 4.09 (1.70 - 9.87) | 0.002 |
| DBP | | | | |
| <90 | 1.00 | | 1.00 | |
| <70 | 2.16 (0.93 - 5.02) | 0.074 | 4.72 (1.69 - 13.12) | 0.003 |
| <50 | 2.56 (1.07 - 6.12) | 0.035 | 4.99 (1.72 - 14.48) | 0.003 |
| Anti-emetics | | | | |
| Yes | 1.00 | | 1.00 | |
| No | 0.64 (0.39 - 1.03) | 0.063 | 1.15 (0.60 - 2.20) | 0.673 |
| Opioids | | | | |
| Yes | 1.00 | | 1.00 | |
| No | 1.52 (0.99 - 2.33) | 0.057 | 1.38 (0.81 - 2.38) | 0.239 |
| Type of feeds | | | | |
| Solids | 1.00 | | 1.00 | |
| Semi-solids | 1.98 (1.17 - 3.36) | 0.012 | 2.08 (1.05 - 4.15) | 0.037 |
| Liquids | 1.06 (0.63 - 1.79) | 0.824 | 1.68 (0.75 - 3.73) | 0.206 |